CLINICAL TRIAL: NCT07400601
Title: A Clinical Cohort Registry Study on Primary PCI for Acute Myocardial Infarction at Zhongshan Hospital
Acronym: ZSPPCI
Status: Recruiting | Type: Observational
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Principal Investigator, Chunfeng Dai, Principal Investigator, Shanghai Zhongshan Hospital
Other Study IDs: B2021-833
Record Dates: First submitted 2026-01-25; First posted 2026-02-10 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-01

CONDITIONS: Acute Myocardial Infarction (AMI)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples Without DNA — All patients will have 5 ml of peripheral venous blood drawn for biochemical analysis before the primary PCI and again on the first day after the procedure.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- AMI patients undergoing primary PCI: Acute myocardial infarction patients undergoing primary PCI
  Interventions: Other: Collection of baseline characteristics

INTERVENTIONS:
Other: Collection of baseline characteristics — Collection of baseline clinical characteristics, procedural details, laboratory results, and medication records

SUMMARY:
This study is a registry-based cohort investigation, prospectively enrolling patients who were diagnosed with acute myocardial infarction and underwent primary percutaneous coronary intervention (PCI) at Zhongshan Hospital, Fudan University, between January 1, 2009, and December 31, 2028. Baseline clinical characteristics, procedural details, laboratory results, and medication records will be systematically collected and documented. The clinical follow-up will encompass both in-hospital monitoring and post-discharge surveillance extending up to two years after the procedure.

DETAILED DESCRIPTION:
This is a registered prospective study that consecutively enrolled patients who were diagnosed with acute myocardial infarction (AMI) and underwent primary percutaneous coronary intervention (PCI) at Zhongshan Hospital, Fudan University, from January 2009 to December 2028. The study recorded each patient's baseline demographics, clinical history, physical examination data, laboratory results, medication usage, and procedural details. The predefined clinical endpoints include both in-hospital and long-term follow-up events. The former encompasses major adverse cardiovascular and cerebrovascular events (MACCE) composed of all-cause death, recurrent myocardial infarction, ischemia-driven repeat revascularization, malignant arrhythmias, acute heart failure, cardiogenic shock, and cerebrovascular accidents, as well as various bleeding events, gout flares, and intraoperative microcirculatory perfusion status during PCI. The latter includes MACCE composed of all-cause death, recurrent myocardial infarction, ischemia-driven repeat revascularization, readmission for acute heart failure, and cerebrovascular accidents, as well as changes in cardiac function during long-term follow-up. The occurrence of malignant tumors was designated as a falsification endpoint to assess the potential impact of confounding factors.

ELIGIBILITY:
Inclusion Criteria:

* Elevated or decreasing levels of cardiac troponin T, with at least one measurement exceeding 0.014 ng/mL;
* Presence of at least one of the following: symptoms of myocardial ischemia; newly onset ischemic changes on ECG; pathological Q wave; imaging evidence of new loss of viable myocardium or regional wall motion abnormalities consistent with ischemia; coronary angiography confirming the presence of a thrombus;
* Undergoing primary PCI;
* Voluntary informed consent to participate in the study.

Exclusion Criteria:

* Inability to complete emergent PCI (e.g., due to intraoperative complications or inability to tolerate the procedure).
* Prior administration of thrombolytic therapy before PCI.
* Diagnosis of type 2 or type 3 myocardial infarction.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study is a registry-based cohort investigation, prospectively enrolling patients who were diagnosed with acute myocardial infarction and underwent primary percutaneous coronary intervention (PCI) at Zhongshan Hospital, Fudan University, between January 1, 2009, and December 31, 2028.
Sampling Method: Non-Probability Sample
Enrollment: 6000 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of MACCE during hospitalization | Periprocedural
  Major adverse cardiovascular and cerebrovascular events (MACCE) occurring during hospitalization, including all-cause death, recurrent myocardial infarction, ischemia-driven repeat revascularization, malignant arrhythmias, acute heart failure, cardiogenic shock, and cerebrovascular accidents
Incidence of MACCE during long-term follow-up | 2 years after PCI
  Major adverse cardiovascular and cerebrovascular events (MACCE) occurring during out-of-hospital follow-up, including all-cause death, recurrent acute myocardial infarction, ischemia-driven repeat revascularization, rehospitalization for acute heart failure, and cerebrovascular accident.

SECONDARY OUTCOMES:
Incidence of bleeding events during hospitalization | Periprocedural
  Various bleeding events during hospitalization
Incidence of gout flare during hospitalization | Periprocedural
  Gout flare during hospitalization
Incidence of myocardial perfusion impairment during primary PCI | Periprocedural
  TIMI < 3

OTHER OUTCOMES:
Cardiac function status during long-term follow-up | up to 2 years
  Document the changes in left ventricular ejection fraction (LVEF) during long-term follow-up. A normal LVEF is over 53%, while an LVEF <50% indicates impaired cardiac systolic function.
The Incidence of Malignant Tumors | 2 years after PCI
  The Incidence of Malignant Tumors During Long-Term Follow-Up

CONTACTS AND LOCATIONS:
Overall Officials: Chunfeng Dai, M.D., Principal Investigator — Fudan University
Locations (1):
- Shanghai Zhongshan Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No
The research involves some confidential content